CLINICAL TRIAL: NCT01398254
Title: The Safety and Efficacy of Femoral Access Versus Radial for Primary Percutaneous Coronary Intervention in ST-Elevation Myocardial Infarction (SAFARI-STEMI Trial)
Brief Title: Femoral Versus Radial Access for Primary PCI
Acronym: SAFARI-STEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Michel Le May, Director of Regional ACS Programs, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MRL-SS; 2011311-01H
Record Dates: First submitted 2011-07-13; First posted 2011-07-20 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Myocardial Infarction; STEMI
Keywords: ST-Elevation Myocardial Infarction; Mortality
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRA (Other): Transradial Access
  Interventions: Procedure: Primary Percutaneous Coronary Intervention (PPCI)
- TFA (Other): Transfemoral Access
  Interventions: Procedure: Primary Percutaneous Coronary Intervention (PPCI)

INTERVENTIONS:
Procedure: Primary Percutaneous Coronary Intervention (PPCI) — Participants will be randomly assigned an access site, radial or femoral, for PPCI.

SUMMARY:
Primary percutaneous coronary intervention (PPCI) has become the dominant strategy for the treatment of ST-elevation myocardial infarction (STEMI), as studies have shown that PPCI is superior to fibrinolytic therapy. Recent evidence suggests that transradial access (TRA) is superior to transfemoral (TFA) for patients undergoing PPCI. Two large trials report a mortality benefit favouring TRA. The results of these two trials could significantly impact practice guidelines and lead to a recommendation that the approach of choice for primary PCI be radial rather than femoral. This would have significant implications for both PCI centers and interventionalists associated with a large impact on practice and education. Yet, many centers and interventionalists in Canada and in the USA prefer TFA and currently feel pressured in making the change to TRA. With that said, these trials did not include new pharmacotherapy and new technology that would likely have closed or eliminated the gap between TFA and TRA by improving the safety and efficacy of these two approaches. Furthermore, these trials were not powered to conclusively show a mortality benefit. The authors of the two large trials emphasized the need for further trials to confirm the benefits of TRA.

The SAFARI-STEMI trial aims to compare TFA with TRA in patients undergoing primary percutaneous intervention (PPCI). The primary outcome will be defined as all cause mortality measured at 30 days. The trial will also evaluate: 1) bleeding events and 2) the composite of death, reinfarction, or stroke defined as major adverse clinical events (MACE). The trial will include the use of antithrombotic therapy with monotherapy, with either bivalirudin or unfractionated heparin; the use of glycoprotein inhibitors IIb/IIIa inhibitors will be avoided. The study will encourage liberal use of vascular closing devices. The trial will also compare delays to reperfusion between the two strategies. Finally, a cost analysis is proposed.

In view of recent publications, there is now a need for a large randomized trial using contemporary adjunct therapies to assess the safety and efficacy of the TRA vs. the TFA in PPCI. The proposed trial aims to conclusively show whether there is a survival benefit associated with the TRA approach.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic chest discomfort of greater or equal to 30 minutes duration,
2. Onset of chest pain of greater or equal to 12 hrs prior to entry into the study,
3. ST segment elevation of > 1 mm (0.1 mV) in two or more contiguous electrocardiographic leads (on a standard 12 lead ECG) or left bundle branch block not known to be old

Exclusion Criteria:

1. Age < 18 yrs
2. Active bleeding
3. Inadequate vascular access from the femoral arteries (i.e. severe peripheral vascular artery disease precluding right or left femoral approach)
4. Abnormal Allen's test precluding either right or left radial approach
5. PCI within the last 30 days
6. Fibrinolytic agents within the last 7 days
7. Warfarin, dabigatran or other oral anticoagulant within the last 7 days
8. Known coagulation disorder (i.e. INR >2.0, platelets <100,000 / mm3)
9. Allergy to aspirin
10. Participation in a study with another investigational device or drug < four weeks
11. Known severe renal impairment (creatinine >200 umol/L)*
12. Known severe contrast (dye) allergy
13. Prior coronary artery bypass surgery
14. Inability to provide informed consent

    * Bivalirudin is contraindicated in renal failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2292 (Actual)
Dates: Start 2011-07; Primary Completion 2018-12 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 days
  The primary outcomes will be all-cause mortality measured at 30 days.

SECONDARY OUTCOMES:
Death, reinfarction, or stroke | 30 days and 6 months
All-cause mortality | 6 months
Reinfarction | 30 days and 6 months
Stroke | 30 days and 6 months
Stent thrombosis | 30 days and 6 months
Bleeding | 30 days
Number of blood transfusions | 30 days
Cardiogenic shock | 30 days
Critical time intervals (including door-to-balloon time) | Index hospitalization
Fluoroscopy time and radiation exposure | Index Catheterization
Length of Hospital Stay | Index hospitalization
Resource utilization | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michel R Le May, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (5):
- Canada (5):
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Center, Thunder Bay, Ontario

REFERENCES:
- [Derived] Marbach JA, Wells G, Santo PD, So D, Chong AY, Russo J, Labinaz M, Dick A, Froeschl M, Glover C, Hibbert B, Marquis JF, MacDougall A, Kass M, Paddock V, Quraishi AUR, Chandrasekhar J, Ghosh N, Bernick J, Le May M. Acute kidney injury after radial or femoral artery access in ST-segment elevation myocardial infarction: AKI-SAFARI. Am Heart J. 2021 Apr;234:12-22. doi: 10.1016/j.ahj.2020.12.019. Epub 2021 Jan 7. PMID 33422518
- [Derived] Le May M, Wells G, So D, Chong AY, Dick A, Froeschl M, Glover C, Hibbert B, Marquis JF, Blondeau M, Osborne C, MacDougall A, Kass M, Paddock V, Quraishi A, Labinaz M. Safety and Efficacy of Femoral Access vs Radial Access in ST-Segment Elevation Myocardial Infarction: The SAFARI-STEMI Randomized Clinical Trial. JAMA Cardiol. 2020 Feb 1;5(2):126-134. doi: 10.1001/jamacardio.2019.4852. PMID 31895439